CLINICAL TRIAL: NCT04735783
Title: Effect of the Perception of Breakfast Consumption on Appetite and Energy Intake in Healthy Males
Brief Title: Placebo Breakfast Consumption, Appetite and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Principal Investigator, Tommy Slater, Principle Investigator, Nottingham Trent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TS_Placebo_2019
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: Breakfast skipping; Energy intake; Energy balance; Appetite hormones; Placebo feeding
MeSH Terms: conditions — Obesity; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake three dietary conditions in a randomised order with at least a four day period in between trials.
Who Masked: Participant
Masking Description: Due to the obvious differences between the three breakfasts meals (viscous, jelly-like placebo breakfast, typical whole-food breakfast, water-only control), participants will be aware that the three trials are different. However, they will not be told that the placebo breakfast contains nearly no energy, and therefore, are blinded to this aspect of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Very low-energy, viscous placebo breakfast (Experimental): Participants will consumed a viscous breakfast meal from a standard bowl with a standard spoon. The volume of the meal will be 5 mL/kg body mass, consisting of 15% (0.75 mL/kg body mass) low-energy flavoured squash, with the remainder made up of tap water. To thicken the solution and increase the perception of energy intake, 0.1 g/kg xanthan gum (a soluble fibre often used as a low-energy thickening agent) will be added and the mixture will be blended thoroughly. An additional 3 mL/kg tap water will be consumed as a drink alongside the meal in this trial.
  Interventions: Dietary Supplement: Placebo breakfast
- Typical, whole-food breakfast (Active Comparator): Participants will consume a standardised meal consisting of puffed rice cereal, semi-skimmed milk, white bread, seedless strawberry jam, and apple juice. This meal will provide 20% of estimated energy requirements, determined by multiplying estimated resting metabolic rate by a physical activity level of 1.6. A measured volume of tap water will be consumed alongside this meal, in order to match total water content of the typical whole-food breakfast to the very low-energy, viscous placebo breakfast.
  Interventions: Dietary Supplement: Typical whole-food breakfast
- Water-only control (Active Comparator): Participants will consume 8 mL/kg body mass of plain tap water to match the total water content of the typical whole-food breakfast and the very low-energy, viscous placebo breakfast.
  Interventions: Dietary Supplement: Water-only control

INTERVENTIONS:
Dietary Supplement: Placebo breakfast — Participants will consume a very low-energy, placebo breakfast meal, but will be unaware of its near complete absence of energy until the end of the study.
  Arms: Very low-energy, viscous placebo breakfast
Dietary Supplement: Typical whole-food breakfast — Participants will consume a typical whole-food breakfast meal, equating to 20% of estimated energy requirements.
  Arms: Typical, whole-food breakfast
Dietary Supplement: Water-only control — Participants will consume a volume of plain water to match the water content of the very low-energy placebo breakfast and the typical whole-food breakfast.
  Arms: Water-only control

SUMMARY:
The purpose of this study was to examine the effects of a very low-energy, viscous placebo breakfast meal on subjective appetite sensations during the morning, and food intake at lunch, compared to a typical whole-food breakfast meal and a water-only control. Participants will not be told that the placebo breakfast contains nearly no energy until the end of the study. The breakfasts will be provided in a randomised order, with a period of at least four days separating the trials. Blood samples will be taken before and after the breakfast is eaten to see how appetite-regulating proteins and blood sugars respond during the morning. Appetite questionnaires will also be completed throughout the morning, and a pasta-based lunch meal will be provided so that voluntary food intake can be measured.

DETAILED DESCRIPTION:
Obesity is a risk factor for several chronic diseases, including type-2 diabetes, heart disease and some forms of cancer. There is clear evidence demonstrating that weight gain occurs progressively over the lifespan, highlighting that preventative action should be taken by young, lean individuals, who may yet develop overweight or obesity later in life. A positive energy imbalance, in which energy intake exceeds energy expenditure for a sustained duration, is known to be the underlying systematic cause of obesity. Therefore, reducing daily energy intake is a seemingly simple solution to the this problem. However, compensatory alterations in appetite regulation which stimulate an increase in energy intake often impede the long-term success of such interventions.

Extending the overnight fasting period, thereby restricting the time available for food intake, has emerged as an effective dietary strategy for reducing daily energy intake and may assist with weight management. Laboratory studies have shown that skipping breakfast typically results in increased appetite during the morning, and an increase in energy intake at lunch. Therefore, the long-term success of skipping breakfast may be reduced by elevated appetite sensations. A recent study which aimed to assess the effects of a very-low energy, placebo breakfast on resistance exercise performance noted that appetite was suppressed after consuming the placebo, despite its lack of energy content. Whether this suppression of appetite following placebo breakfast consumption results in a reduced energy intake at lunch, is currently unknown. Therefore, the investigators are interested to examine the subjective and hormonal appetite responses to placebo breakfast consumption, compared with these responses to an overt breakfast consumption trial an overt breakfast skipping trial, and whether these changes result in any differences in voluntary energy intake at lunch.

The present study is a randomised, controlled, crossover study in which fourteen healthy, habitual breakfast-consuming (self-reported) males will consume a very low-energy, viscous placebo breakfast, a typically consumed, whole-food breakfast, and a water-only control. At least four days will separate trials.

Participants will firstly complete a pre-screening session in which anthropometric data will be collected. This will be used to determine the energy content of the typical whole-food breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker.
* Habitually consuming breakfast at least 3 days per week.
* Have maintained a stable weight for 6 months (self-reported).
* No known history of gastric, digestive, cardiovascular or renal disease.

Exclusion Criteria:

* Food allergies, dislike or intolerance of study foods or drinks.
* Not currently on a weight management program or have irregular eating patterns (i.e. extended fasting periods >8h other than overnight - self reported).
* Use of medication that may affect hormone concentrations.
* Excessive alcohol consumption (>4 units/day).
* Intensive training schedule (>10 hours/week).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Voluntary energy intake (Kilocalories) at a laboratory-based test lunch meal | 195 minutes post-breakfast provision.
  A laboratory-based meal consisting of pasta, tomato sauce and olive oil will be provided to participants in excess of expected consumption. Participants will be permitted 20 minutes to eat as much or as little as they desire, until 'comfortably full and satisfied'.

SECONDARY OUTCOMES:
Visual Analogue Scale for Subjective Ratings of Appetite | Baseline, 10 minutes, 30 minutes, 60 minutes, 120 minutes, 195 minutes, 215 minutes, 275 minutes post-breakfast provision.
  Time-course of subjective ratings of hunger between breakfast provision and one hour after consuming lunch, measured using an appetite visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, desire to eat and prospective food consumption. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Acylated ghrelin | Baseline, 60 minutes, 180 minutes post-breakfast provision.
  Time-course of acylated ghrelin plasma concentrations across experimental trials.
Peptide tyrosine-tyrosine (PYY) | Baseline, 60 minutes, 180 minutes post-breakfast provision.
  Time-course of PYY plasma concentrations across experimental trials.
Blood glucose concentration | Baseline, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes post-breakfast provision.
  Time-course of blood glucose concentrations across experimental trials.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Loughborough University, Loughborough
  - Nottingham Trent University, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naharudin MN, Adams J, Richardson H, Thomson T, Oxinou C, Marshall C, Clayton DJ, Mears SA, Yusof A, Hulston CJ, James LJ. Viscous placebo and carbohydrate breakfasts similarly decrease appetite and increase resistance exercise performance compared with a control breakfast in trained males. Br J Nutr. 2020 Mar 16:1-9. doi: 10.1017/S0007114520001002. Online ahead of print. PMID 32174286
- [Background] Mears SA, Dickinson K, Bergin-Taylor K, Dee R, Kay J, James LJ. Perception of Breakfast Ingestion Enhances High-Intensity Cycling Performance. Int J Sports Physiol Perform. 2018 Apr 1;13(4):504-509. doi: 10.1123/ijspp.2017-0318. Epub 2018 May 14. PMID 28952831
- [Background] Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Effect of extended morning fasting upon ad libitum lunch intake and associated metabolic and hormonal responses in obese adults. Int J Obes (Lond). 2016 Feb;40(2):305-11. doi: 10.1038/ijo.2015.154. Epub 2015 Aug 17. PMID 26278005
- [Background] Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Carbohydrate-rich breakfast attenuates glycaemic, insulinaemic and ghrelin response to ad libitum lunch relative to morning fasting in lean adults. Br J Nutr. 2015 Jul 14;114(1):98-107. doi: 10.1017/S0007114515001506. Epub 2015 May 25. PMID 26004166
- [Background] Clayton DJ, Barutcu A, Machin C, Stensel DJ, James LJ. Effect of Breakfast Omission on Energy Intake and Evening Exercise Performance. Med Sci Sports Exerc. 2015 Dec;47(12):2645-52. doi: 10.1249/MSS.0000000000000702. PMID 25970668
- [Background] Betts JA, Chowdhury EA, Gonzalez JT, Richardson JD, Tsintzas K, Thompson D. Is breakfast the most important meal of the day? Proc Nutr Soc. 2016 Nov;75(4):464-474. doi: 10.1017/S0029665116000318. Epub 2016 Jun 13. PMID 27292940
- [Background] Clayton DJ, James LJ. The effect of breakfast on appetite regulation, energy balance and exercise performance. Proc Nutr Soc. 2016 Aug;75(3):319-27. doi: 10.1017/S0029665115004243. Epub 2015 Dec 14. PMID 26653842
- [Background] Astbury NM, Taylor MA, Macdonald IA. Breakfast consumption affects appetite, energy intake, and the metabolic and endocrine responses to foods consumed later in the day in male habitual breakfast eaters. J Nutr. 2011 Jul;141(7):1381-9. doi: 10.3945/jn.110.128645. Epub 2011 May 11. PMID 21562233
- [Background] Levitsky DA, Pacanowski CR. Effect of skipping breakfast on subsequent energy intake. Physiol Behav. 2013 Jul 2;119:9-16. doi: 10.1016/j.physbeh.2013.05.006. Epub 2013 May 11. PMID 23672851
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233
- [Derived] Slater T, Mode WJA, Hough J, James RM, Sale C, James LJ, Clayton DJ. Effect of the perception of breakfast consumption on subsequent appetite and energy intake in healthy males. Eur J Nutr. 2022 Apr;61(3):1319-1330. doi: 10.1007/s00394-021-02727-5. Epub 2021 Nov 11. PMID 34766208